CLINICAL TRIAL: NCT06141564
Title: Molecular and Immunological Signatures in Recurrent Hepatocellular Carcinoma (HCC)
Brief Title: Detect and Expunge Concealed Tumors of the Liver
Acronym: DTECT-Liver
Status: Active, not recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: 108 Military Central Hospital, Hanoi, Viet Nam (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB00389479
Record Dates: First submitted 2023-11-14; First posted 2023-11-21 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, liver cancer tissues and non-cancerous tissues
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Early stage HCC
- Compensated cirrhosis
- Chronic hepatitis without cirrhosis

SUMMARY:
The investigators long-term goal is to identify molecular and immunological signatures that can be used as biomarkers to accurately predict early recurrence and inform immunotherapeutic strategies in patients with hepatocellular carcinoma (HCC) after hepatectomy. As an initial step toward this long-term investigation, represented by this proposal, the investigators aim to comprehensively and globally describe the patterns of autoantibody expressions, the possible role in disease outcomes, and the relationship between these autoantibodies to tumor-specific/tumor-associated antigens by histologic examination as well as to peripheral immune characteristics in HCC patients with or without recurrence after surgery.

DETAILED DESCRIPTION:
The current methods for early detection and therapy for recurrent HCC are generally ineffective and mostly inaccessible to patients worldwide. Thus, there is an urgent unmet medical need to have a sensitive and accessible method for monitoring and guiding therapeutic strategy for HCC recurrence, which will improve the prognosis of patients.

The investigators current understanding of the mechanisms underpinning the onset and progression of HCC recurrence is incomplete. While tumor-related factors, including tumor size, number and differentiation, and underlying liver disease, are known risk factors for recurrence following curative therapies; evidence suggests that the recurrent mechanism is also governed by complex, poorly understood host immune responses. Tumor- and liver-infiltrating immune cells on the progression and recurrence of HCC have been documented. Tumor-infiltrating lymphocytes are believed to inhibit tumor growth, improving the prognosis of human malignancies. Inflammatory cytokines, including members of the interleukin (IL) and IL-11, contribute to hepatocyte proliferation and are also associated with cancer development after surgery. Unlike primary HCC, relapsed tumors have a higher immune evasion characteristic due to the accumulation of inhibitory cytokines and molecules. Moreover, the tumor microenvironment also plays a key role in the recurrence of HCC. Many immunosuppressive mechanisms, such as increased regulatory T cells and myeloid-derived suppressor cells with decreased cytotoxic T cells, are implicated in HCC recurrence.

Identifying panels of tumor antigens that elicit a humoral response may have utility in cancer screening, diagnosis, or prognosis. Such antigens may also have utility in designing immunotherapy against the disease. A proteomic-based approach for identifying tumor antigens that induce autoantibodies to tumor antigens can be detected using the Human Proteome (HuProt) arrays. The HuProt arrays, comprising 21,154 unique full-length proteins can be deployed to survey serum autoantibodies using primary or recurrent HCC samples. Likewise, profiling peripheral immune cell populations and cytokines will add another dimension to the landscape of HCC recurrence and host immune modulation.

In summary, identifying novel molecular and immunological markers in circulation and/or cancerous tissues is desirable to predict the risk of early primary and recurrent HCCs. This, coupled with several promising forms of immunotherapy for HCC that are currently available can help guide future therapies for HCCs.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Collection of biosamples at baseline (sera, liver cancer and non liver cancer tissues, Peripheral blood mononuclear cells (PBMCs)) each of the 3-month interval follow ups (serum and PBMCs) for a total of 4 during the study follow up duration 1 year post-hepatectomy.
* Early-stage HCC eligible for hepatectomy for curative intention. Early HCC (Stage A) is limited to a single tumor <5 cm in diameter or three tumors that are each <3cm.
* Stated willingness to comply with all study procedures and availability for the duration of the study and up to 3 years post-study follow up
* Adults aged 18 or older
* Both genders and all ethnicities
* Willingness to give written, informed consent to be enrolled into the study database
* Reside in Vietnam at the time of study and provides contact information (email and/or cell phone number for texting)
* No prior or current treatment of HCC
* No cancer history within 5 years
* No participation in other trial for HCC Treatment
* No significant hepatic decompensation
* No hepatorenal syndrome
* Alpha fetoprotein (AFP) test labs within 90 days irrespective of AFP titer
* Two phone numbers and personal identification numbers (CMND number)
* No known AIDS related diseases
* No significant co-morbid conditions with life expectancy <2 years

Exclusion Criteria:

* Individuals who cannot, do not want to, or refused to sign the informed consent form (ICF)
* Any serious or active medical or psychiatric illness, which, in the opinion of the investigator, would interfere with patient treatment, assessment or compliance with the protocol
* Documentation was not adequate
* Known HIV positive
* Taking immunosuppressants
* Having any autoimmune diseases based on clinical and/or laboratory availabilities

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Early stage HCCs who are eligible for hepatectomy Cirrhosis due to any etiologies, MELD <= 15 Chronic hepatitis due to any etiologies, without cirrhosis or HCC
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
HCC recurrence diagnosed by dynamic contrast enhanced CT | Post-hepatectomy up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Doan Dao, MD, Principal Investigator — Johns Hopkins School of Medicine; Binh T Mai, MD, PhD, Principal Investigator — 108 Military Central Hospital, Hanoi, Viet Nam; Chi V Dang, MD, PhD, Principal Investigator — Johns Hopkins University; Heng Zhu, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- 108 Military Central Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No